CLINICAL TRIAL: NCT00818870
Title: A Randomized, Open-Label, Cross-Over, Dose-Ranging Study to Assess the Effect of Vecam 40/300 and Vecam 20/300 Administered at Bedtime Compared to Omeprazole 20 mg Administered Before Breakfast on Gastric pH
Brief Title: Effect of Vecam 40/300 and Vecam 20/300 Compared to Omeprazole 20 mg on Gastric pH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vecta Ltd. (Industry)
Responsible Party: Richard E. Lowenthal, Vecta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCT006
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; GERD; Nocturnal GERD; Heartburn; Nighttime Heartburn; Nocturnal Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omeprazole 20 mg (Active Comparator)
  Interventions: Drug: Omeprazole
- Vecam 20/300 (Experimental)
  Interventions: Drug: Vecam
- Vecam 40/300 (Experimental)
  Interventions: Drug: Vecam

INTERVENTIONS:
Drug: Omeprazole — 20 mg capsule, orally, once daily (before breakfast) for 5 days.
  Arms: Omeprazole 20 mg
Drug: Vecam — 1 capsule, orally, once daily at bedtime for 5 days.
  Arms: Vecam 20/300
Drug: Vecam — 1 capsule, orally, once daily at bedtime for 5 days.
  Arms: Vecam 40/300

SUMMARY:
The study is designed to assess and compare the effect of Vecam 40/300, Vecam 20/300 and Omeprazole 20 mg (a standard FDA approved GERD treatment) on the control of gastric pH.

DETAILED DESCRIPTION:
Eligible H. pylori negative, normal gastric acid secreting, healthy volunteers will be treated by the study medications in a randomized, open-label, cross-over study.Up to 60 volunteers may be enrolled to ensure that at least 30 subjects will complete all the study treatments. Omeprazole 20 mg will be administered before breakfast. Vecam 40/300 and Vecam 20/300 will be administered at bedtime w/o food. 24-hour gastric pH will be measured after the fifth dose (day 5).Following screening procedures, subjects will be randomly assigned to receive the different treatments.

All pH measurements will be done in the study center under supervised conditions. All drug administrations will be supervised.

This study is part of the Vecam clinical development plan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, H. pylori negative status (by Urea Breath Test)
* Male or female subjects
* Age 18-55 years
* Able to tolerate the placement of a nasogastric pH probe at screening
* Baseline Gastric pH≤2
* Use of acceptable form of birth control in females with child-bearing potential
* Had not used any form of tobacco (e.g. smoking or chewing) for the last year
* Can swallow a size "00" capsule without difficulty
* Willing to comply with study protocol
* Signed Informed Consent form

Exclusion Criteria:

* BMI > 40
* Slow or poor Omeprazole metabolizers (heterozygous or homozygous, respectively) based on CYP2C19 genotyping test.
* Any significant history of / or concurrent gastrointestinal diseases or conditions such as:

  * GERD
  * Acute gastrointestinal bleeding
  * Zollinger Ellison Syndrome or Gastric hypersecretory condition
  * Known Barrett's esophagus
  * Esophageal stricture
  * Peptic ulcer disease (gastric or duodenal) or family history of peptic ulcer disease
  * Gastric outlet obstruction
  * Gastroparesis
* Significant medical history or concurrent illness as determined by the principal investigator
* Any medical disorder that alters the normal gastric acid secretion profile as determined by the principal investigator
* History of diabetes mellitus
* Significant laboratory abnormalities as determined by the principal investigator
* Known metabolic alkalosis, hypocalcemia, sodium restricted diet, hypokalemia, respiratory alkalosis
* Pregnant or lactating women
* Had been treated with any investigational drug or therapy or participated in a clinical trial within 30 days prior to entering the trial
* Use of any medication other than contraception or hormone replacement therapy; OTC drugs other than vitamins or occasional acetaminophen within 30 days prior to entering the trial or during the trial
* Use of NSAID medications within 30 days prior to entering the trial (e.g. Ibuprofen, Aspirin, Naproxen etc)
* Positive urine test for alcohol or other drugs
* Concurrent use of gastric anti-secretory drugs such as defined below:

  * Use of a PPI 30 days prior to each stage or during the trial
  * Use of H2RA 14 days prior to each stage or during the trial
  * Concurrent use of antacids (including over-the-counter) 24 hours prior to each stage or during the trial
* Use of any medication that modifies gastric acid secretion 30 days prior to or during the trial.
* Had ingested grapefruit within 14 days of dose administration in any trial period
* Significant drug allergy or known hypersensitivity to any of the ingredients in the trial drugs Omeprazole, Succinic Acid or to Lidocaine
* Consumption of coffee within 48 hours of dose administration in any trial period.
* Had donated blood within 30 days of entering the trial
* Known positive serology for HBV, HCV or HIV
* Any reason which makes the subject a poor candidate based on the physician's discretion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess whether Vecam 40/300 administered at bedtime w/o food is pharmacodynamically superior to Omeprazole 20 mg administered before breakfast, calculated as percent time gastric pH ≥4 for the 24-hour interval after the fifth dose. | 5 days

SECONDARY OUTCOMES:
To assess whether Vecam 40/300 administered at bedtime w/o food is pharmacodynamically superior to Vecam 20/300 administered at bedtime w/o food calculated as percent time gastric pH ≥4 for the 24-hour interval after the fifth dose. | 5 days
To assess whether Vecam 20/300 administered at bedtime w/o food is pharmacodynamically superior to Omeprazole 20 mg administered before breakfast, calculated as percent time gastric pH ≥4 for the 24-hour interval after the fifth dose. | 5 days
To assess whether Vecam 40/300 administered at bedtime w/o food is pharmacodynamically superior to Vecam 20/300 administered at bedtime w/o food calculated as percent time gastric pH ≥4 during nocturnal hours after the fifth dose. | 5 days
To assess whether Vecam 40/300 administered at bedtime w/o food is pharmacodynamically superior to Omeprazole 20 mg administered before breakfast calculated as percent time gastric pH ≥4 during nocturnal hours after the fifth dose | 5 days
To assess whether Vecam 20/300 administered at bedtime w/o food is pharmacodynamically superior to Omeprazole 20 mg administered before breakfast calculated as percent time gastric pH ≥4 during nocturnal hours after the fifth dose. | 5 days
To asses Vecam 40/300 administered at bedtime w/o food vs. Omeprazole 20 mg administered before breakfast calculated as percent time pH ≥4 during 24-hour interval and nocturnal hours at early dosing days. | 5 days
To assess the safety of Vecam 40/300 and Vecam 20/300 administered at bedtime vs. Omeprazole 20 mg administered before breakfast during treatment period. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Vijayalakshmi S Pratha, MD, Principal Investigator — Clinical Applications Laboratories Inc.
Locations (1):
- Clinical Applications Laboratories Inc., San Diego, California, United States

REFERENCES:
- [Derived] Chowers Y, Atarot T, Pratha VS, Fass R. The effect of once daily omeprazole and succinic acid (VECAM) vs once daily omeprazole on 24-h intragastric pH. Neurogastroenterol Motil. 2012 May;24(5):426-31, e208-9. doi: 10.1111/j.1365-2982.2012.01884.x. Epub 2012 Feb 28. PMID 22372795